CLINICAL TRIAL: NCT00563706
Title: A Randomized, Double-Blind, Placebo-Controlled, Risperidone-Referenced, Parallel-Group, Adaptive-Design Study of the Efficacy, Safety, and Tolerability of Vabicaserin (SCA-136) in Subjects With Acute Exacerbations of Schizophrenia
Brief Title: Study Evaluating Vabicaserin in Subjects With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3153A1-2203; B1911032
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Results first posted 2014-03-20 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — vabicaserin; Risperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: vabicaserin
- 2 (Active Comparator): 4mg/day
  Interventions: Drug: risperidone
- 3 (Placebo Comparator): matching placebo
  Interventions: Other: placebo

INTERVENTIONS:
Drug: vabicaserin — This study will utilize a randomized, double-blind, placebo-controlled, comparator-referenced, multicenter, parallel-group adaptive design with placebo, risperidone (4 mg/day), and up to 7 treatment arms of vabicaserin (50, 100, 150, 200, 300, 400 and 600 mg/day) over the course of the study
  Arms: 1
Drug: risperidone
  Arms: 2
Other: placebo
  Arms: 3

SUMMARY:
The primary purpose of this protocol is to establish the efficacy, safety, and tolerability of vabicaserin (SCA-136) using a once a day capsule in subjects with acute exacerbations of schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy, men and women, aged 18 to 65.
* Hospitalization because of an acute exacerbation of schizophrenia with a diagnosis of schizophrenia established greater than 1 year.
* Ability to remain hospitalized for the duration of the screening period and for 4 weeks of double-blind treatment.

Exclusion Criteria:

* Current Axis I primary psychiatric diagnosis other than schizophrenia (DSM-IV-TR criteria).
* Current diagnosis or history of substance abuse or dependence (DSM-IV-TR criteria), including alcohol (except for nicotine), within 3 months before baseline (day -1).
* Subjects taking high or chronic doses of benzodiazepine at the screening evaluation who, in the investigator's judgment, would be likely to have severe withdrawal symptoms upon discontinuation.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2007-12; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (31):
- United States (30):
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Cerritos, California
  - Pfizer Investigational Site, Escondido, California
  - Pfizer Investigational Site, Garden Grove, California
  - Pfizer Investigational Site, Glendale, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Torrance, California
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Aventura, Florida
  - Pfizer Investigational Site, Hollywood, Florida
  - Pfizer Investigational Site, Kissimmee, Florida
  - Pfizer Investigational Site, Hoffman Estates, Illinois
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Lake Charles, Louisiana
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Rockville, Maryland
  - Pfizer Investigational Site, Hamilton, New Jersey
  - Pfizer Investigational Site, Willingboro, New Jersey
  - Pfizer Investigational Site, Cedarhurst, New York
  - Pfizer Investigational Site, Holliswood, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Butner, North Carolina
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Bellaire, Texas
  - Pfizer Investigational Site, DeSoto, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Arlington, Virginia
  - Pfizer Investigational Site, Portsmouth, Virginia
- Pfizer Investigational Site, Kingston, Ontario, Canada

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3153A1-2203&StudyName=Study%20Evaluating%20Vabicaserin%20in%20Subjects%20With%20Schizophrenia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 204 participants were randomized, of which 202 participants received at least 1 dose of double-blind test article.
Groups:
- Placebo: Four placebo capsules matched to vabicaserin (SCA-136) orally once daily up to Day 28 during double-blind (DB) treatment phase followed by 2 placebo capsules matched to vabicaserin orally once daily up to Day 35 during taper phase.
- Vabicaserin 50 mg: One vabicaserin 50 milligram (mg) capsule and 3 placebo capsules matched to vabicaserin (equivalent to vabicaserin 50 mg) orally once daily up to Day 28 during double-blind treatment phase followed by 2 placebo capsules matched to vabicaserin orally once daily up to Day 35 during taper phase.
- Vabicaserin 100 mg: One vabicaserin 100 mg capsule and 3 placebo capsules matched to vabicaserin (equivalent to vabicaserin 100 mg) orally once daily up to Day 28 during double-blind treatment phase followed by 2 placebo capsules matched to vabicaserin orally once daily up to Day 35 during taper phase.
- Vabicaserin 150 mg: One vabicaserin 50 mg capsule, 1 vabicaserin 100 mg capsule, and 2 placebo capsules matched to vabicaserin (equivalent to vabicaserin 150 mg) orally once daily up to Day 28 during double-blind treatment phase followed by 1 vabicaserin 50 mg capsule and 1 placebo capsule matched to vabicaserin (equivalent to vabicaserin 50 mg) orally once daily up to Day 32 and then 2 placebo capsules matched to vabicaserin orally once daily up to Day 35 during taper phase.
- Vabicaserin 200 mg: Two vabicaserin 100 mg capsules and 2 placebo capsules matched to vabicaserin (equivalent to vabicaserin 200 mg) orally once daily up to Day 28 during double-blind treatment phase followed by 1 vabicaserin 100 mg capsule and 1 placebo capsule matched to vabicaserin (equivalent to vabicaserin 100 mg) orally once daily up to Day 32 and then 1 vabicaserin 50 mg capsule and 1 placebo capsule matched to vabicaserin (equivalent to vabicaserin 50 mg) orally once daily up to Day 35 during taper phase.
- Vabicaserin 300 mg: Three vabicaserin 100 mg capsules and 1 placebo capsule matched to vabicaserin (equivalent to vabicaserin 300 mg) orally once daily up to Day 28 during double-blind treatment phase followed by 1 vabicaserin 100 mg capsule and 1 placebo capsule matched to vabicaserin (equivalent to vabicaserin 100 mg) orally once daily up to Day 32 and then 1 vabicaserin 50 mg capsule and 1 placebo capsule matched to vabicaserin (equivalent to vabicaserin 50 mg) orally once daily up to Day 35 during taper phase.
- Vabicaserin 400 mg: Two vabicaserin 200 mg capsules and 2 placebo capsules matched to vabicaserin (equivalent to vabicaserin 400 mg) orally once daily up to Day 28 during double-blind treatment phase followed by 1 vabicaserin 200 mg capsule and 1 placebo capsule matched to vabicaserin (equivalent to vabicaserin 200 mg) orally once daily up to Day 32 and then 1 vabicaserin 100 mg capsule and 1 placebo capsule matched to vabicaserin (equivalent to vabicaserin 100 mg) orally once daily up to Day 35 during taper phase.
- Vabicaserin 600 mg: Three vabicaserin 200 mg capsules and 1 placebo capsule matched to vabicaserin (equivalent to vabicaserin 600 mg) orally once daily up to Day 28 during double-blind treatment phase followed by 1 vabicaserin 200 mg capsule and 1 placebo capsule matched to vabicaserin (equivalent to vabicaserin 200 mg) orally once daily up to Day 32 and then 1 vabicaserin 100 mg capsule and 1 placebo capsule matched to vabicaserin (equivalent to vabicaserin 100 mg) orally once daily up to Day 35 during taper phase.
- Risperidone: One risperidone 4 mg capsule and 3 placebo capsules matched to risperidone (equivalent to risperidone 4 mg) orally once daily up to Day 28 during double-blind treatment phase followed by 1 risperidone 2 mg capsule and 1 placebo capsule matched to risperidone (equivalent to risperidone 2 mg) orally once daily up to Day 35 during taper phase.
Period: DB Treatment Period (Day 1 up to Day 28)
Arm/Group | Placebo | Vabicaserin 50 mg | Vabicaserin 100 mg | Vabicaserin 150 mg | Vabicaserin 200 mg | Vabicaserin 300 mg | Vabicaserin 400 mg | Vabicaserin 600 mg | Risperidone
Started | 37 | 18 | 8 | 19 | 16 | 19 | 12 | 30 | 43
Completed | 20 | 13 | 3 | 9 | 11 | 14 | 9 | 16 | 32
Not Completed | 17 | 5 | 5 | 10 | 5 | 5 | 3 | 14 | 11
Not completed — Adverse Event | 4 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 5
Not completed — Lack of Efficacy | 2 | 1 | 2 | 4 | 1 | 2 | 2 | 5 | 1
Not completed — Withdrawal by Subject | 9 | 3 | 2 | 5 | 4 | 3 | 1 | 6 | 3
Not completed — Discontinuation of Study by Sponsor | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Period: Taper Phase (Day 29 up to Day 35)
Arm/Group | Placebo | Vabicaserin 50 mg | Vabicaserin 100 mg | Vabicaserin 150 mg | Vabicaserin 200 mg | Vabicaserin 300 mg | Vabicaserin 400 mg | Vabicaserin 600 mg | Risperidone
Started | 20 | 13 | 3 | 9 | 11 | 14 | 9 | 16 | 32
Completed | 20 | 13 | 3 | 9 | 11 | 14 | 9 | 16 | 32
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized participants who received at least 1 dose of double-blind test article.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Vabicaserin 50 mg | Vabicaserin 100 mg | Vabicaserin 150 mg | Vabicaserin 200 mg | Vabicaserin 300 mg | Vabicaserin 400 mg | Vabicaserin 600 mg | Risperidone | Total
Number analyzed (Participants) | 37 | 18 | 8 | 19 | 16 | 19 | 12 | 30 | 43 | 202
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.05 (9.88) | 43.22 (10.17) | 41.25 (4.89) | 40.53 (11.43) | 42.94 (8.27) | 40.74 (10.29) | 38.17 (9.73) | 43.60 (9.25) | 42.72 (9.93) | 42.07 (9.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 1 | 4 | 5 | 3 | 0 | 6 | 10 | 41
  Male | 29 | 14 | 7 | 15 | 11 | 16 | 12 | 24 | 33 | 161

OUTCOME MEASURES:

1. Primary Outcome: Positive and Negative Symptom Scale (PANSS) Total Score at Baseline
Description: PANSS assesses the positive symptoms, negative symptoms, and general psychopathology specifically associated with schizophrenia. The scale consists of 30 items. Each item is rated on a scale from 1 (symptom not present) to 7 (symptoms extremely severe). The sum of the 30 items is defined as the PANSS total score and ranges from 30 to 210; higher score indicates greater severity.
Time Frame: Baseline
Population: Modified intent-to-treat (mITT) population included all randomized participants who received at least 1 dose of double-blind test article, had baseline and at least 1 on-therapy PANSS total score.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Vabicaserin 50 mg | Vabicaserin 100 mg | Vabicaserin 150 mg | Vabicaserin 200 mg | Vabicaserin 300 mg | Vabicaserin 400 mg | Vabicaserin 600 mg | Risperidone
Number analyzed (Participants) | 35 | 17 | 8 | 18 | 16 | 18 | 12 | 28 | 42
units on a scale | 94.74 (11.18) | 94.24 (8.42) | 96.88 (14.54) | 101.33 (12.97) | 93.06 (8.84) | 94.39 (8.73) | 92.83 (10.25) | 95.54 (12.46) | 91.43 (10.83)

2. Primary Outcome: Change From Baseline in Positive and Negative Symptom Scale (PANSS) Total Score at Day 28
Description: as for outcome 1
Time Frame: Baseline, Day 28
Population: mITT population included all randomized participants who received at least 1 dose of double-blind test article, had baseline and at least 1 on-therapy PANSS total score. Here "N" (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vabicaserin 50 mg | Vabicaserin 100 mg | Vabicaserin 150 mg | Vabicaserin 200 mg | Vabicaserin 300 mg | Vabicaserin 400 mg | Vabicaserin 600 mg | Risperidone
Number analyzed (Participants) | 21 | 13 | 3 | 10 | 11 | 14 | 9 | 17 | 32
units on a scale | -17.03 (3.59) | -4.72 (4.87) | -10.26 (8.35) | -5.41 (5.18) | -13.42 (5.17) | -6.13 (4.80) | -13.84 (5.93) | -7.30 (4.09) | -15.59 (3.20)
Statistical Analysis 1: Comparison: Placebo vs Vabicaserin 50 mg; Mixed effects model was used to assess the treatment effects with change in PANSS total score from baseline as response variable, treatment, visit, and treatment by visit as fixed factors and baseline value as a covariate; Test type: Superiority or Other; p = 0.043, Mixed Models Analysis; Least Squares (LS) Mean Difference = -12.30, 95% CI 2-sided [-24.24 to -0.37]
Statistical Analysis 2: Comparison: Placebo vs Vabicaserin 100 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.457, Mixed Models Analysis; LS Mean Difference = -6.77, 95% CI 2-sided [-24.70 to 11.16]
Statistical Analysis 3: Comparison: Placebo vs Vabicaserin 150 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.067, Mixed Models Analysis; LS Mean Difference = -11.61, 95% CI 2-sided [-24.03 to 0.81]
Statistical Analysis 4: Comparison: Placebo vs Vabicaserin 200 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.567, Mixed Models Analysis; LS Mean Difference = -3.61, 95% CI 2-sided [-16.02 to 8.80]
Statistical Analysis 5: Comparison: Placebo vs Vabicaserin 300 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.070, Mixed Models Analysis; LS Mean Difference = -10.90, 95% CI 2-sided [-22.71 to 0.92]
Statistical Analysis 6: Comparison: Placebo vs Vabicaserin 400 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.647, Mixed Models Analysis; LS Mean Difference = -3.18, 95% CI 2-sided [-16.87 to 10.50]
Statistical Analysis 7: Comparison: Placebo vs Vabicaserin 600 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.075, Mixed Models Analysis; LS Mean Difference = -9.73, 95% CI 2-sided [-20.46 to 1.00]
Statistical Analysis 8: Comparison: Placebo vs Risperidone; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.765, Mixed Models Analysis; LS Mean Difference = -1.44, 95% CI 2-sided [-10.92 to 8.04]

3. Secondary Outcome: Positive and Negative Symptom Scale (PANSS) Positive Subscale Score
Description: PANSS positive subscale assesses positive symptoms associated with schizophrenia. The positive subscale consists of 7 items (delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution, and hostility). Each item is rated on a scale from 1 (symptom not present) to 7 (symptoms extremely severe). Total positive subscale scores range from 7 to 49; higher score indicates greater severity.
Time Frame: Baseline, Day 7, 14, 21, 28
Population: Because of the failure of all vabicaserin doses to meet the primary efficacy objective, the study was terminated prematurely and planned analyses of secondary efficacy endpoints were not performed.
Arm/Group | Placebo | Vabicaserin 50 mg | Vabicaserin 100 mg | Vabicaserin 150 mg | Vabicaserin 200 mg | Vabicaserin 300 mg | Vabicaserin 400 mg | Vabicaserin 600 mg | Risperidone
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Positive and Negative Symptom Scale (PANSS) Negative Subscale Score
Description: PANSS negative subscale assesses negative symptoms associated with schizophrenia. The negative subscale consists of 7 items (blunted affect, emotional withdrawal, poor rapport, passive/apathetic social withdrawal, difficulty in abstract thinking, lack of spontaneity and flow of conversation, and stereotyped thinking). Each item is rated on a scale from 1 (symptom not present) to 7 (symptoms extremely severe). Total negative subscale scores range from 7 to 49; higher score indicates greater severity.
Time Frame: Baseline, Day 7, 14, 21, 28
Population: as for outcome 3
Arm/Group | Placebo | Vabicaserin 50 mg | Vabicaserin 100 mg | Vabicaserin 150 mg | Vabicaserin 200 mg | Vabicaserin 300 mg | Vabicaserin 400 mg | Vabicaserin 600 mg | Risperidone
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Positive and Negative Symptom Scale (PANSS) General Psychopathology Subscale Score
Description: General psychopathology subscale assesses general psychopathology symptoms associated with schizophrenia. The general psychopathology subscale consists of 16 items (somatic concern, anxiety, guilt feelings, tension, mannerisms/posturing, depression, motor retardation, uncooperativeness, unusual thought content, disoriented, poor attention, lack of judgment/insight, disturbance of volition, poor impulse control, preoccupation, and active social avoidance). Each item is rated on a scale from 1 (symptom not present) to 7 (symptoms extremely severe). Total general psychopathology subscale scores range from 16 to 112; higher score indicates greater severity.
Time Frame: Baseline, Day 7, 14, 21, 28
Population: as for outcome 3
Arm/Group | Placebo | Vabicaserin 50 mg | Vabicaserin 100 mg | Vabicaserin 150 mg | Vabicaserin 200 mg | Vabicaserin 300 mg | Vabicaserin 400 mg | Vabicaserin 600 mg | Risperidone
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Positive and Negative Symptom Scale (PANSS) Cognition Cluster Subscale Score
Description: Cognition cluster subscale assesses cognitive symptoms associated with schizophrenia. The cognition cluster subscale score is a sum of 5 items from positive, negative and general psychopathology subscales (conceptual disorganization, difficulty in abstract thinking, poor attention, lack of judgment and insight, and preoccupation). Each item is rated on a scale from 1 (symptom not present) to 7 (symptoms extremely severe). Total cognition cluster subscale scores range from 5 to 35; higher score indicates greater severity.
Time Frame: Baseline, Day 7, 14, 21, 28
Population: as for outcome 3
Arm/Group | Placebo | Vabicaserin 50 mg | Vabicaserin 100 mg | Vabicaserin 150 mg | Vabicaserin 200 mg | Vabicaserin 300 mg | Vabicaserin 400 mg | Vabicaserin 600 mg | Risperidone
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Percentage of Participants With Response As Per Positive and Negative Symptom Scale (PANSS) Total Score
Description: Responders were defined as 20 percent (%) responders and 50 % responders. A 20% responder was a participant whose PANSS total score was decreased by at least 20% from baseline to the week of assessment. A 50% responder was a participant whose PANSS total score was decreased by at least 50 % from baseline to the week of assessment. PANSS total score assesses the positive symptoms, negative symptoms, and general psychopathology specifically associated with schizophrenia. The scale consists of 30 items. Each item is rated on a scale from 1 (symptom not present) to 7 (symptoms extremely severe). The sum of the 30 items is defined as the PANSS total score and ranges from 30 to 210; higher score indicates greater severity.
Time Frame: Baseline, Day 7, 14, 21, 28
Population: as for outcome 3
Arm/Group | Placebo | Vabicaserin 50 mg | Vabicaserin 100 mg | Vabicaserin 150 mg | Vabicaserin 200 mg | Vabicaserin 300 mg | Vabicaserin 400 mg | Vabicaserin 600 mg | Risperidone
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Clinical Global Impression - Severity (CGI-S) Score
Description: CGI-S: 7-point clinician rated scale to assess severity of participant's current illness state; range: 1 (normal - not ill at all) to 7 (among the most extremely ill patients).
Time Frame: Baseline, Day 7, 14, 21, 28
Population: as for outcome 3
Arm/Group | Placebo | Vabicaserin 50 mg | Vabicaserin 100 mg | Vabicaserin 150 mg | Vabicaserin 200 mg | Vabicaserin 300 mg | Vabicaserin 400 mg | Vabicaserin 600 mg | Risperidone
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Clinical Global Impression - Improvement (CGI-I) Score
Description: CGI-I: 7-point clinician rated scale to assess global improvement in the participant's clinical state compared to baseline; range: 1 (very much improved) to 7 (very much worse).
Time Frame: Day 7, 14, 21, 28
Population: as for outcome 3
Arm/Group | Placebo | Vabicaserin 50 mg | Vabicaserin 100 mg | Vabicaserin 150 mg | Vabicaserin 200 mg | Vabicaserin 300 mg | Vabicaserin 400 mg | Vabicaserin 600 mg | Risperidone
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Calgary Depression Scale for Schizophrenia (CDSS) Score
Description: CDSS: 9-item clinician rated scale, validated for rating the severity of depressive symptoms in participants with schizophrenia. Each item is rated on a 4-point scale ranging from 0 (absent) to 3 (severe). CDSS total score is the sum of each item scores and ranges from 0 to 27; higher score indicates more severity of symptoms.
Time Frame: Baseline, Day 7, 14, 21, 28
Population: as for outcome 3
Arm/Group | Placebo | Vabicaserin 50 mg | Vabicaserin 100 mg | Vabicaserin 150 mg | Vabicaserin 200 mg | Vabicaserin 300 mg | Vabicaserin 400 mg | Vabicaserin 600 mg | Risperidone
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Placebo | Vabicaserin 50 mg | Vabicaserin 100 mg | Vabicaserin 150 mg | Vabicaserin 200 mg | Vabicaserin 300 mg | Vabicaserin 400 mg | Vabicaserin 600 mg | Risperidone
Serious Adverse Events (participants affected / at risk) | 4/37 | 0/18 | 1/8 | 0/19 | 0/16 | 1/19 | 2/12 | 2/30 | 3/43
Other Adverse Events (participants affected / at risk) | 28/37 | 12/18 | 6/8 | 11/19 | 13/16 | 13/19 | 10/12 | 23/30 | 35/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=37) | Vabicaserin 50 mg (N=18) | Vabicaserin 100 mg (N=8) | Vabicaserin 150 mg (N=19) | Vabicaserin 200 mg (N=16) | Vabicaserin 300 mg (N=19) | Vabicaserin 400 mg (N=12) | Vabicaserin 600 mg (N=30) | Risperidone (N=43)
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Homicidal ideation (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intentional self-injury (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Schizophrenia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Schizophrenia, undifferentiated type (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=37) | Vabicaserin 50 mg (N=18) | Vabicaserin 100 mg (N=8) | Vabicaserin 150 mg (N=19) | Vabicaserin 200 mg (N=16) | Vabicaserin 300 mg (N=19) | Vabicaserin 400 mg (N=12) | Vabicaserin 600 mg (N=30) | Risperidone (N=43)
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gaze palsy (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Anal pruritus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 4 | 3
Diarrhoea (Gastrointestinal disorders) | 5 | 2 | 0 | 1 | 2 | 1 | 0 | 2 | 3
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 3
Dyspepsia (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 1 | 1 | 2 | 1 | 1 | 2 | 3 | 4
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Stomach discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 3
Toothache (Gastrointestinal disorders) | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 4
Vomiting (Gastrointestinal disorders) | 2 | 2 | 1 | 0 | 0 | 1 | 2 | 3 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Pain (General disorders) | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pitting oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 1
Sluggishness (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sexually transmitted disease (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Medical device complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 2 | 1
Hepatic enzyme increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 1 | 1 | 0 | 1 | 0 | 1 | 2 | 0 | 6
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Akathisia (Nervous system disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3
Choreoathetosis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 1 | 0 | 2 | 0 | 1 | 5 | 3
Drooling (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Dyskinesia (Nervous system disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Extrapyramidal disorder (Nervous system disorders) | 3 | 1 | 1 | 3 | 2 | 0 | 0 | 2 | 3
Headache (Nervous system disorders) | 5 | 1 | 1 | 1 | 1 | 1 | 1 | 3 | 4
Lethargy (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sedation (Nervous system disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 2
Sinus headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 4
Tardive dyskinesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 1
Agitation (Psychiatric disorders) | 3 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 1 | 2
Bruxism (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Nightmare (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Paranoia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 2 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0 | 2 | 1 | 0 | 1
Schizophrenia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Galactorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 2
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Because of the failure of all vabicaserin doses to meet the primary efficacy objective, the study was terminated prematurely and planned analyses of secondary efficacy endpoints were not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.